CLINICAL TRIAL: NCT06263907
Title: Preemptive Efficacy of Stellate Ganglion Block for Prevention of Post Mastectomy Depression
Brief Title: Stellate Ganglion Block for Prevention of Post Mastectomy Depression
Acronym: SGB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anaesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: stellate ganglion block
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Mastectomy; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomization into two equal groups using computer-generated random numbers prior to surgery of 70 each; Group S: will receive ipsilateral stellate gangalion block and Group C: will receive no block.
Who Masked: Participant, Investigator
Masking Description: The anesthesiologist, who will be responsible for opening the envelope and do the block or not according to the group besides, evaluation of its success and covering the skin over the site of ipsilateral stellate gangalion with sterile dressing in both groups, will not be involved in data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate gangalion block group (Group S) (Experimental): Patients will receive ipsilateral stellate gangalion block (4ml) bupivacaine 0.25 %+( 4ml) normal saline + (8mg) dexamethasone in a total 10 ml
  Interventions: Procedure: Stellate gangalion block
- Control group (Group C) (No Intervention): Patients will not receive stellate gangalion block

INTERVENTIONS:
Procedure: Stellate gangalion block — The efficacy of Preoperative ipsilateral stellate gangalion block on the occurrence of postmastectomy depression and pain compared with no block
  Arms: Stellate gangalion block group (Group S)

SUMMARY:
Complications after mastectomy include chronic pain and depression.

DETAILED DESCRIPTION:
A mastectomy is surgery could be associated with complications include chronic pain and depression. In female breast cancer patients, the incidence of postoperative depression was 46.55%. Stellate ganglion block had been used for treating post-traumatic stress disorder (PTSD) and depression symptoms even in its prevention. Also, it used in treatment of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age ranging from 18 to 65 years
* American Society of Anesthesiologists (ASA) no more than II
* Had unilateral cancer breast
* Scheduled to do unilateral modified radical mastectomy

Exclusion Criteria:

* Pregnant female
* Existing Horner syndrome
* Had any neuromuscular disease
* Had allergy to local anesthetics
* History of use of analgesics
* Had any deformity or a previous surgery in the neck or ipsilateral arm or breast
* Had any contraindication to the procedure (coagulation disorders, local infection, sepsis)
* Had any contraindication to the sympathetic blockade (decompensate cardiopulmonary or hemodynamic disorders)
* History of psychotic disorder including depression, bipolar disorder or personality disorder
* Patient with Beck Depression Inventory (BDI) score more than 13

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients scheduled to do unilateral modified radical mastectomy
Enrollment: 140 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of postmastectomy depression | 6 months postoperatively
  Beck Depression Inventory (BDI) score

SECONDARY OUTCOMES:
incidence of postmastectomy depression | 3 months postoperatively
  Beck Depression Inventory (BDI) score
the need for postoperative antidepressant | during the first 6 months postoperatively
  needed or not
acute postoperative pain at the incision site (breast and the axilla) | every 12 hour for the first 48 hour recorded
  Numerical rating scale (NRS) (0-10)
chronic postmastectomy pain at the incision site | at 3 and 6 months postoperatively
  Numerical rating scale (NRS) (0-10)
incidence of nausea and vomiting | during first 3 postoperative days
  occurred or not
Functional pain in the ipsilateral shoulder | during the first 6 months postoperatively
  extended from the shoulder to the elbow or to the hand either associated with swelling, changing in the colour or temperature of that limb or associated with reduction in the range of the movement (elbow extension or arm abduction or fixed flexion deformity
Any complications related to stellate ganglion injection | within 1 day postoperatively
  local hematoma, persistent postoperative horner's syndrome or respiratory distress

CONTACTS AND LOCATIONS:
Locations (1):
- Maha, Al Mansurah, Egypt